CLINICAL TRIAL: NCT01736488
Title: A Randomized, Double-Blind, Phase IV Clinical Study to Evaluate the Antihypertensive Efficacy and Changes of Neurohormonal Markers of Fimasartan and Atenolol With Exaggerated Blood Pressure Response During Exercise in Essential Hypertensive Patients
Brief Title: Clinical Study to Evaluate the Antihypertensive Efficacy and Changes of Neurohormonal Markers of Fimasartan and Atenolol With Exaggerated Blood Pressure Response During Exercise in Essential Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FA-CT-401
Record Dates: First submitted 2012-11-19; First posted 2012-11-29 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Hypertension; Antihypertensive efficacy; Neurohormonal markers; Blood Pressure Response; Exercise
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — fimasartan; Atenolol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fimasartan 60mg (Experimental): 60mg/day of Fimasartan will be oral administered for the study period (8 weeks)
  Interventions: Drug: Fimasartan
- Atenolol 50mg (Active Comparator): 50mg/day of Atenolol will be oral administered for the study period (8 weeks)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Fimasartan — Fimasartan 60mg
  Other Names: Kanarb
  Arms: Fimasartan 60mg
Drug: Atenolol — Atenolol 50mg
  Other Names: Tenolmin
  Arms: Atenolol 50mg

SUMMARY:
The purpose of this study is to evaluate the antihypertensive efficacy and changes of neurohormonal markers of fimasartan and atenolol with exaggerated blood pressure response during exercise in essential hypertensive patients.

DETAILED DESCRIPTION:
After subjects have signed informed consent voluntarily, when they are taking hypertension medication, they go through screening period for 7 days including wash-out period.

After screening and wash-out period, subjects take the placebo for 14 days (Maximum 21 days), and evaluate their suitability to Inclusion and Exclusion criteria.

Patients, who evaluated the proper subject for this clinical trial, are allocated to experimental group (Fimasartan 60mg) or Control group (Atenolol 50mg) randomly at a ratio 1:1 and their investigational drugs will be administered daily for the study period (8 weeks). Subjects visit their investigators twice during treatment period, when they take their investigational drugs for 4 weeks, and 8 weeks.

The placebo period will be single-blinded and the treatment allocation in this study will be double-blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who agreed to participate in this clinical trial and submitted the written informed consent
2. Subjects aged 20 to 75 years
3. Essential hypertension patients who are measured more 140mmHg, less than 170mmHg of sitting systolic blood pressure(SiSBP) or more 90mmHg, less than 110mmHg of sitting diastolic blood pressure(SiDBP) at baseline(Day 0)
4. men who are measured more 210mmHg, women who are measured more 190mmHg or increasing more than 50mmHg after exercise at baseline(Day 0)
5. Subject who considered to understand this clinical trial, be cooperative,and able to be followed-up whole of the clinical trial period

Exclusion Criteria:

1. Patients who are measured the difference of mean blood pressure of one arm under sitting diastolic blood pressure(SiDBP) 10mmHg or SiSBP 20mmHg at screening and baseline visit
2. more 170mmHg of mean Sitting systolic blood pressure(SiSBP)or more 110mmHg of mean Sitting diastolic blood pressure(SiDBP) before exercise at baseline(Day 0)
3. Patients with secondary hypertension
4. Patients with orthostatic hypotension who has sign and symptom
5. Patients with severe insulin dependent or uncontrolled diabetes mellitus (HbA1c>9, regimen change of oral hypoglycemic agent, using insulin)
6. Patients with severe heart disease, ischemic heart disease within 6 months, peripheral vascular disease, Percutaneous transluminal coronary angiography(PTCA), Coronary artery bypass graft(CABG)
7. Patients with significant ventricular tachycardia, atrial fibrillation, atrial flutter or other significant arrhythmia
8. Patients with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve disease
9. Patients with severe cerebrovascular disease
10. Patients with known severe or malignancy retinopathy
11. Patients with wasting disease, autoimmune disease, connective tissue disease at present and/or previous
12. Patients with significant investigations; abnormal renal function (Creatinine more 1.5 times than upper limit of normal), abnormal liver function(AST, ALT more 2 times than upper limit of normal), severe fatty liver disease needed medication
13. Patients with surgical and medical disease that is able to be affect to absorption, distribution, metabolism and excretion
14. Patients who have a story or evidence of alcohol or drug abuse within 2 years
15. Childbearing and breast-feeding women
16. Female who plan to become pregnancy or have a possibility of pregnancy but don't prevent conception with acknowledged methods
17. Patients with Bronchial Asthma
18. Patients expected to live less than 1 year with tumor or chronic disease
19. Patients with hepatitis B or C
20. Patients with history of allergic reaction to any angiotensin II antagonist
21. Patients who took medicine within 12 weeks from screening visit or is going on the progress of other clinical trial
22. Subject who are judged unsuitable to participate in this clinical trial by investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The difference of sitting Systolic Blood Pressure(SiSBP) between at the peak compared to at resting | After 8 weeks from baseline visit
  To compare the difference of sitting Systolic Blood Pressure(SiSBP) at the peak compared to at resting between Fimasartan 60mg group and Atenolol 50mg group

SECONDARY OUTCOMES:
The difference of sitting Diastolic Blood Pressure(SiDBP) at the peak compared to at resting | After 8 weeks from baseline visit
  To compare the difference of sitting Diastolic Blood Pressure(SiDBP), Heart Rate, Neurohormonal markers at the peak compared to at resting between Fimasartan 60mg group and Atenolol 50mg group
The difference of sitting Systolic Blood Pressure(SiSBP) at each exercising stage compared to at resting | After 8 weeks from baseline visit
  To compare the difference of sitting Systolic Blood Pressure(SiSBP), sitting Diastolic Blood Pressure(SiDBP), Heart Rate at each exercising stage and at recovery compared to at resting between Fimasartan 60mg group and Atenolol 50mg group
The difference of sitting Systolic Blood Pressure(SiSBP) among at resting, each exercising stage and recovery | After 8 weeks from baseline visit
  To compare the difference of sitting Systolic Blood Pressure(SiSBP), sitting Diastolic Blood Pressure(SiDBP), Heart Rate, neurohormonal markers among at resting, each exercising stage and recovery between Fimasartan 60mg group and Atenolol 50mg group

CONTACTS AND LOCATIONS:
Overall Officials: Jong Won Ha, PhD, Principal Investigator — Yonsei University
Locations (4):
- South Korea (4):
  - Hallym University Medical Center, Anyang
  - Gachon University Gil Hospital, Incheon
  - Severance Hospital, Seoul
  - Kangnam Severance Hospital, Seoul